CLINICAL TRIAL: NCT03615820
Title: Propolis-based Nanovesicles as Oromuco-adhesive Film: Novel Therapeutic Drug Delivery System for Treatment of Oral Recurrent Aphthous Ulcer
Brief Title: Niosomal Propolis as Oromucoadhesive Film: In-vitro, Ex-vivo & In-vivo Investigations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Mona Gamal Mohamed Afifi Arafa, Lecturer, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPEADHNIO-2018-4
Record Dates: First submitted 2018-03-30; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Drug Effect; Drug Effect Prolonged
Keywords: Nanovesicles; Aphthous ulcer
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Intervention Model Description: Volunteers will be divided into two groups; each group contained 12 volunteers who will receive one formula of the selected formulae
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Niosomal PPE oromucoadhesive film (Experimental): Niosomal PPE oromucoadhesive film in which PPE entrapped in niosomes then incorporated in oromucoadhesive films
  Interventions: Drug: Niosomal PPE oromucoadhesive film; Drug: Oromucoadhesive film
- Oromucoadhesive film (Placebo Comparator): Oromucoadhesive film that has no niosomal PPE in its content
  Interventions: Drug: Niosomal PPE oromucoadhesive film; Drug: Oromucoadhesive film

INTERVENTIONS:
Drug: Niosomal PPE oromucoadhesive film — Niosomal PPE oromucoadhesive film in which Propolis entrapped in niosomal vesicles and incorporated in oromucoadhesive film
Drug: Oromucoadhesive film — Oromucoadhesive film without PPE control testing which represents Placebo group

SUMMARY:
A total of 24 patients suffering from RAU, they were divided into two groups each included 12 patients. The first group was treated by the propolis mucoadhesive film and the second group received the film without the active component (placebo group).Patients were handed a checklist for monitoring the actual improvement of the clinical parameters which included; duration of disappearance of pain after film application (hours), duration of complete healing of the aphthous ulcer (weeks), onset of ulcer size reduction after film application (days), duration of propolis film adherence onto the oral mucosa (hours) and finally the level of patient satisfaction scaled from 1-10.

DETAILED DESCRIPTION:
The present study have been performed on a total of 24 patients suffering from RAU, they were divided into two groups each included 12 patients. The first group was treated by the propolis mucoadhesive film and the second group received the film without the active component (placebo group). Patients were recruited from the out-patient clinic of the Faculty of Dentistry, British University in Egypt during a period of 6 months.

Patients were subjected to thorough clinical examination and history obtaining in order to diagnose the oral ulcer by an oral medicine specialist, they were thoroughly informed about the study and only those with the oral ulcer within the first day to the third day of appearance were included in the present study.

The exclusion criteria in the present study were the presence of systemic or local disease such as hepatitis, cardiac conditions, hypertension, diabetes mellitus, renal problems, mental disorders, AIDS and also the use of any immunosuppressive drugs or systemic corticosteroids during last three months or using steroid treatment locally in last month, also any nutritional supplements, folic acid or antioxidants, pregnancy and nursing.

All patients were asked to avoid using antiseptics, antibiotics or analgesics, during the study as they might aid in curing the oral ulcers. Patients were blinded of receiving either propolis or placebo. They were warned about the potentiality of allergic responses that could happen to some people and that in case of occurrence of such side effect immediate termination of using the film should be implemented.

The patients were first instructed how to apply the mucoadhesive film of 2 cm2 on the oral ulcer and pasted by applying a light force with the finger tip for 20 s, and then were asked to apply it two times per day and to refrain from eating for at least one hour after the film application on the oral ulcer.

Patients were handed a checklist for monitoring the actual improvement of the clinical parameters which included; duration of disappearance of pain after film application (hours), duration of complete healing of the aphthous ulcer (weeks), onset of ulcer size reduction after film application (days), duration of propolis film adherence onto the oral mucosa (hours) and finally the level of patient satisfaction scaled from 1-10. After total healing of the oral RAU, checklists were recollected from patients, the results were tabulated and statistical analysis were conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffer from aphthous ulcer

Exclusion Criteria:

* Chronic diseases ,
* Hospitalized

Ages: 40 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Determination of the onset of ulcer size reduction | Fifteen Days
  Niosomal PPE in oromuco-adhesive film was prepared & given to 12 patients to examine the onset of ulcer size reduction The patients were first instructed how to apply the mucoadhesive film of 2 cm2 on the oral ulcer and then they were handed a checklist for monitoring the actual improvement that was indicated by the reduction of the size of ulcer.

SECONDARY OUTCOMES:
Duration of complete ulcer healing | Fifteen Days
  oromuco-adhesive film was prepared & given to 12 patients to examine the duration of complete healing.The patients were first instructed how to apply the mucoadhesive film of 2 cm2 on the oral ulcer and then they were handed a checklist for monitoring the actual improvement that was indicated by the complete healing of ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Mona G Arafa, PhD, Principal Investigator — The British University in Egypt
Locations (2):
- Egypt (2):
  - Mona G Arafa, New Cairo, Cairo Governorate
  - Mona G Arafa, Cairo